CLINICAL TRIAL: NCT05225532
Title: CardioneuROablation: coMparison of Right Versus Left Atrial Approach in Patients With Reflex syNcope. The Roman 2 Randomized Controlled Prospective Study
Brief Title: Cardioneuroablation: Comparison of Right Versus Left Atrial Approach in Patients With Reflex Syncope
Acronym: ROMAN2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant differences between the groups were noted during interim analysis (as scheduled in the protocol) and the study was stopped because the final result was obtained
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Professor, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 89/2021
Record Dates: First submitted 2021-12-28; First posted 2022-02-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Reflex Syncope
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LA group (Experimental): Patients randomized to procedure performed in the left atrium
  Interventions: Other: Radiofrequency ablation
- RA group (Active Comparator): Patients randomized to procedure performed in the right atrium
  Interventions: Other: Radiofrequency ablation

INTERVENTIONS:
Other: Radiofrequency ablation — Radiofrequency ablation of ganglionated plexi located in the left or right atrium

SUMMARY:
Introduction. Reflex vaso-vagal syncope (VVS) is the most frequent cause of transient loss of consciousness and it's treatment remains a challenge. Cardioneuroablation (CNA) is a relatively new and promising method, however, the optimal technique for performing CNA has not been established.

Aim. To compare effectiveness of CNA performed in the right atrium (RA) versus left atrium (LA) in achieving total vagal denervation and in preventing syncope recurrences.

Methods. Study group. Consecutive patients with recurrent cardioinhibitory or mixed VVS, undergoing CNA between January 2022 and February 2024 will be randomized to the RA or LA groups.

CNA is performed under general anesthesia with muscle relaxation using a 3.5 mm irrigated tip contact force catheter and ablation index.The whole procedure is performed under intracardiac echocardiography (ICE) guidance. Efficacy of vagal denervation is assessed using extracardiac vagal stimulation (ECVS). Before starting RF delivery baseline electrophysiological parameters are measured. Next, baseline ECVS from the left and right jugular veins is performed.

In the LA group, after gaining transseptal access under ICE guidance, an electroanatomical map of the LA is created and anatomically-based ablation of GP from the LA is performed. Firstly, septal GP are ablated and if total vagal denervation is not achieved, GP located close to left pulmonary veins are ablated. If ECVS still shows vagal response, additional RF applications are delivered in the RA. Then, final ECVS is performed and procedure is finished.

In the RA group, GP located in this chamber are ablated and if ECVS shows persistent vagal response, transseptal puncture is performed and ablation in the LA is performed. Afterwards, final ECVS is performed.

Duration of follow-up is two years. Patients will attend check-up visits at 3, 12 and 24 months with standard ECG, 24hr ambulatory ECG and QoL assessment.

Primary endpoint is complete vagal denervation measured by ECVS (no sinus arrest and no AVB after CNA) using LA approach only versus RA approach only Secondary endpoints include final ECVS results and follow-up data - syncope/presyncope recurrences and QoL.

DETAILED DESCRIPTION:
Introduction. Reflex vaso-vagal syncope (VVS) is the most frequent cause of transient loss of consciousness in general population. It markedly decreases quality of life and may lead to injury. The mechanisms of VVS are complex with enhanced parasympathetic activity being one of the most important, leading to prolonged asystole and/or vasodilatation and syncope.

Treatment of VVS remains a challenge. Non-pharmacological treatment such as fluid and salt intake, avoiding situations triggering syncope or tilt training is not effective in a significant proportion of subjects with syncope. Pharmacotherapy is even less effective. Syncope recurs in 50% of patients. Alternative therapy, especially in patients with prolonged asystole, is pacemaker implantation, recommended by the guidelines in patients aged > 40 years with documented spontaneous cardioinhibitory VVS and severe symptoms. However, permanent pacing occurs ineffective in at least 12-25% of patients. In addition, VVS occurs predominantly in young persons in whom permanent pacing should be avoided as much as possible. Thus, there is a need for new treatment options in VVS.

Cardioneuroablation (CNA) is a relatively new method, introduced by Pachon et al in 2005. To date, numerous small and medium volume reports have been published, showing CNA efficacy between 40% and 100%, at a mean level of around 85-90% at one-year follow-up. The procedure consists of radio-frequency (RF) ablation of ganglionated plexi (GP) located in the epicardial fat around right (RA) and left atrium (LA). The RF-induced injury of GP markedly diminishes vagal tone because, contrary to the adrenergic nerve endings, parasympathetic fibers predominate in GP and do not regenerate, therefore, procedural effects are probably durable.

The optimal technique for performing CNA has not been established and operators use various approaches. There are at least three issues to be addressed. The first one is the choice of cardiac chamber for CNA. Some operators perform RF ablation in the RA only whereas others in both atria or mainly in the LA.

Secondly, the procedural end-points are also inconsistent. Some use simple measures such as increase in heart rate (HR) and changes in other electrophysiological parameters suggesting vagal withdrawal whereas others use extra cardiac vagal stimulation (ECVS) performed from the right (RIJV) and left internal jugular veins (LIJV) to demonstrate sinus arrest and atrio-ventricular (AVB) block at baseline and lack of ECVS effects after successful total vagal denervation. The ECVS was introduced by Pachon and seems to be an excellent intra-procedural end-point, however, it is not clear whereas it's use is required to obtain favorable long-term results. Moreover, it is not known whether total vagal denervation (no sinus arrest and no AVB) is mandatory or maybe partial denervation (no sinus arrest or AVB) is sufficient to prevent syncope recurrences.

Thirdly, methods for identification of GP are imperfect and variable. Ideally, GP should be identified in individual patient using specific markers such as MIBG because there may be inter-patient differences in GP locations. However, these methods are costly, time-consuming, poorly accessible and difficult to merge with electro-anatomical systems (EAM) used during RF ablation. Therefore, other methods such as intracardiac spectral mapping, searching for fractionated potentials or intracardiac high-frequency stimulation has been tried. However, all these methods have their own drawbacks and the majority of operators use simple anatomical approach, sometimes combined with previously mentioned techniques.

In summary, there are many unknowns in CNA. The present project aims to address two of these uncertainties. First, which approach more effectively causes intra-procedural total vagal denervation, and second - which approach is associated with better outcome - simple and faster RA only versus more complex LA ablation.

Aim. To compare effectiveness of RA CNA versus LA CNA in achieving total vagal denervation and in preventing syncope recurrences.

Hypothesis. CNA using RA approach significantly less frequently causes complete vagal denervation and is significantly less effective than LA in prevention of syncope recurrences.

Methods. Study group. Consecutive patients with recurrent cardioinhibitory or mixed VVS, undergoing CNA between January 2022 and February 2024 will be randomized to the RA or LA groups. The institutional Ethics Committee approval was obtained on the 20th of October, 2021, approval number 89/2021.

Cardioneuroablation The procedure is performed under general anesthesia with muscle relaxation using a 3.5 mm irrigated tip catheter (Navistar ThermoCool SmartTouch; Biosense Webster, Diamond Bar, California, USA) with contact force module and electroanatomical system Carto 3 (Biosense Webster, Diamond Bar, California, USA). The quality of RF applications is controlled by ablation index which is set at 450-500 at anterior LA wall, 400-450 at the posterior LA wall and in the RA, and 300-400 in the CS. The whole procedure is performed under intracardiac echocardiography (ICE) guidance (Acuson SC2000 Ultrasound Machine, Siemens, Erlangen, Germany and ACUSON AcuNav™ Ultrasound Catheter, Biosense Webster, Diamond Bar, California, USA). The ECVS is performed using standard diagnostic catheter and neurostimulator designed by Pachon (Sao Paulo, Brazil) which generates pulsed electric field with pulse amplitude of 1 V/kg body weight up to 70 V, 50 ms width, 50 Hz frequency, delivered over 5-8 sec. Before starting RF delivery baseline electrophysiological parameters are measured. Next, baseline ECVS from the left and right jugular veins is performed. The tip of diagnostic catheter is placed as close as possible to the vagus nerve under fluoroscopic and ultrasonographic guidance. This is followed by RF ablation which protocol differs between LA and RA groups. The protocol allows for the extension of the procedure (from RA to LA and from LA to RA) if vagal response during ECVS is be still present after ablation from RA or LA only.

The LA group. After gaining transseptal access under ICE guidance, an electroanatomical map of the LA is created and anatomically-based ablation of GP from the LA is performed. Ablation is started at the site of the anterior right GP (ARGP) and is continued downwards along the anterior part of a common vestibulum of the right pulmonary veins (PV), opposite to the right-sided ablation lesions. Second, area of the right inferior GP (RIGP), close to the RIPV is ablated. At this point ECVS is performed and if there is no vagal response, the procedure is finished. If not, inferior LGP (LIGP) is ablated, ECVS is repeated and the area of left superior GP (LSGP) is ablated if vagal response is still present. If after all these applications ECVS still shows vagal response, further RF applications at the sites of GP located close to the left PV, especially in the grove between LSPV and LA appendage (site of ligament of Marshall), are performed and final ECVS in LA is performed.

If full denervation (asystole or AVB still present at ECVS) after ablation in the LA is not achieved, ablation catheter is moved from LA to RA, and subsequent applications are performed in the RA at the RAGP and RIGP area. The location of phrenic nerve and sinus node area are identified in order to avoid RF applications at these sites. If vagal response using ECVS is still present after this additional set of RF lesions in the RA, sites close to Ao-SVC GP and in the CS are targeted. After that, final ECVS is performed and procedure is finished regardless of ECVS result.

The RA group. In this group, ablation is started from the supero-posterior area targeting RSGP, followed by the infero-posterior area targeting RIGP. The location of phrenic nerve and sinus node area are identified in order to avoid RF applications at these sites. Next, ECVS is performed and if vagal response is still present, sites close to Ao-SVC GP and in the CS are targeted.

If after ablation of all GP sites in the RA the ECVS still shows vagal response, transseptal puncture is performed and ablation is moved to the LA where all GP are ablated as in the LA group. Afterwards, final ECVS is performed and procedure is finished regardless of ECVS result.

Heparin administration. In the LA group, heparin is administered intravenously in a dose of 100 units per kg at the time of transseptal puncture and additional doses are administered during ablation to maintain ACT > 350 sec. In the RA group, heparin is not administered, however, if there is a need to move with ablation to the LA, heparin is given as in the LA group.

Measurements of EP parameters. Standard EP parameters such as heart rate, sinus node recovery time (uncorrected and corrected) as well as atrio-ventricular conduction (Wenckebach point using incremental pacing and atrio-ventricular node refractory period using extrastimulus technique) are measured at baseline and after completion of CNA.

Post-CNA atropine test. At the end of the procedure 2 mg of atropine is administered and sinus rate after 1 and 2 minutes following injection is assessed.

Follow-up. Duration of follow-up is two years. Patients will attend check-up visits at 3, 12 and 24 months with standard ECG, 24hr ambulatory ECG and QoL assessment. Data on syncope and presyncope recurrences will be collected.

Quality of life. Quality of life will be assessed before and 3, 12 and 24 months after CNA using dedicated questionnaire. This questionnaire consists of 9 questions with 6 choices and 3 questions with 5 choices. The overall maximum score is 57. The higher the score the poorer the quality of life is.

Statistical analysis Results will be presented as means ± SD or numbers and percentages. Numeric variables will be compared using the two-sided paired T-student test. A p value of <0.05 will be considered significant.

Calculated sample size. The minimum number of subjects that need to be enrolled in a study in order to have sufficient statistical power to detect a treatment effect is 98 (49 patients in each group) with alfa value of 0.05, beta error of 0.2 and power of 0.8 assuming that complete vagal denervation measured using ECVS will be 75% in the RA group and 95% in the LA group.

Interim Analysis The first interim analysis will be performed after 20 patients recruited into each RA and LA groups. If in at least 10 out of 20 patients randomized to any study group ECVS will continue to show vagal response after CNA performed in a single chamber (RA first or LA first) the study will be stopped and protocol modification will be considered.

ELIGIBILITY:
Inclusion Criteria:

* 1. Documented spontaneous or tilt-induced syncope with at least 3 seconds of asystole due to sinus arrest or AVB, refractory to standard non-pharmacological treatment.
* 2. High syncope burden (> 1 syncope per year or > 3 presyncopal events during preceding 12 months) or very severe syncope in the past, leading to injury.
* 3. Significantly decreased quality of life due to syncope (>20 points in QoL questionnaire dedicated to patients with syncope [17]).
* 4. Standard ECG and 24hr ambulatory ECG recorded within one month before procedure.
* 5. Positive baseline atropine test defined as at least 30% increase in sinus rate compared with baseline value.
* 6. Obtained written informed consent.
* 7. Age > 16 years

Exclusion Criteria:

* 1. Other possible and treatable causes of syncope such as orthostatic hypotension, IST, POTS, significant cardiac disease, cardiac arrhythmia or abnormalities of vertebrobasilar arteries
* 2. History of stroke or TIA
* 3. History of cardiac surgery
* 4. Contraindications to ablation in the right or left atrium

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
No sinus arrest and no AVB after procedure completed in the LA only or RA only | 1 day
  Assessment with the use of ECVS whether complete vagal denervation was achieved after procedure performed in the left atrium only versus right atrium only

SECONDARY OUTCOMES:
No sinus arrest and no AVB at the end of procedure | 1 day
  Assessment with the use of ECVS whether complete vagal denervation was achieved at the end of the whole procedure
Efficacy of CNA - syncope recurrences | 24 months
  Number of patients with syncope recurrence during two-year follow-up
Efficacy of CNA - Time to first syncope recurrence | 1 day - 24 months
  Time to first syncope recurrence
Efficacy of CNA - syncope burden | 24 months
  Syncope burden (number of syncopal episodes during two years)
Efficacy of CNA - presyncope burden | 24 months
  Presyncope burden (number of presyncopal episodes during two years)
Point-scale for quality of life | 24 months
  Quality of life before and after completion the study is assessed using 9 questions with 6 choices and 3 questions with 5 choices. The overall maximum score is 57.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kulakowski, MD PhD, Principal Investigator — Postgraduate Centre for Medical Eductaion
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
raw data will be available on request from other researches when the study is completed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 2024
Access Criteria: personal e-mail contact

REFERENCES:
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM, Leyva F, Linde C, Abdelhamid M, Aboyans V, Arbelo E, Asteggiano R, Baron-Esquivias G, Bauersachs J, Biffi M, Birgersdotter-Green U, Bongiorni MG, Borger MA, Celutkiene J, Cikes M, Daubert JC, Drossart I, Ellenbogen K, Elliott PM, Fabritz L, Falk V, Fauchier L, Fernandez-Aviles F, Foldager D, Gadler F, De Vinuesa PGG, Gorenek B, Guerra JM, Hermann Haugaa K, Hendriks J, Kahan T, Katus HA, Konradi A, Koskinas KC, Law H, Lewis BS, Linker NJ, Lochen ML, Lumens J, Mascherbauer J, Mullens W, Nagy KV, Prescott E, Raatikainen P, Rakisheva A, Reichlin T, Ricci RP, Shlyakhto E, Sitges M, Sousa-Uva M, Sutton R, Suwalski P, Svendsen JH, Touyz RM, Van Gelder IC, Vernooy K, Waltenberger J, Whinnett Z, Witte KK. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Europace. 2022 Jan 4;24(1):71-164. doi: 10.1093/europace/euab232. No abstract available. PMID 34455427
- [Result] Brignole M, Menozzi C, Moya A, Andresen D, Blanc JJ, Krahn AD, Wieling W, Beiras X, Deharo JC, Russo V, Tomaino M, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Pacemaker therapy in patients with neurally mediated syncope and documented asystole: Third International Study on Syncope of Uncertain Etiology (ISSUE-3): a randomized trial. Circulation. 2012 May 29;125(21):2566-71. doi: 10.1161/CIRCULATIONAHA.111.082313. Epub 2012 May 7. PMID 22565936
- [Result] Brignole M, Russo V, Arabia F, Oliveira M, Pedrote A, Aerts A, Rapacciuolo A, Boveda S, Deharo JC, Maglia G, Nigro G, Giacopelli D, Gargaro A, Tomaino M; BioSync CLS trial Investigators. Cardiac pacing in severe recurrent reflex syncope and tilt-induced asystole. Eur Heart J. 2021 Feb 1;42(5):508-516. doi: 10.1093/eurheartj/ehaa936. PMID 33279955
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Result] Yao Y, Shi R, Wong T, Zheng L, Chen W, Yang L, Huang W, Bao J, Zhang S. Endocardial autonomic denervation of the left atrium to treat vasovagal syncope: an early experience in humans. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):279-86. doi: 10.1161/CIRCEP.111.966465. Epub 2012 Jan 24. PMID 22275485
- [Result] Sun W, Zheng L, Qiao Y, Shi R, Hou B, Wu L, Guo J, Zhang S, Yao Y. Catheter Ablation as a Treatment for Vasovagal Syncope: Long-Term Outcome of Endocardial Autonomic Modification of the Left Atrium. J Am Heart Assoc. 2016 Jul 8;5(7):e003471. doi: 10.1161/JAHA.116.003471. PMID 27402231
- [Result] Aksu T, Golcuk E, Yalin K, Guler TE, Erden I. Simplified Cardioneuroablation in the Treatment of Reflex Syncope, Functional AV Block, and Sinus Node Dysfunction. Pacing Clin Electrophysiol. 2016 Jan;39(1):42-53. doi: 10.1111/pace.12756. Epub 2015 Oct 26. PMID 26411271
- [Result] Aksu T, Guler TE, Bozyel S, Yalin K. Selective vagal innervation principles of ganglionated plexi: step-by-step cardioneuroablation in a patient with vasovagal syncope. J Interv Card Electrophysiol. 2021 Apr;60(3):453-458. doi: 10.1007/s10840-020-00757-3. Epub 2020 May 11. PMID 32394104
- [Result] Debruyne P, Rossenbacker T, Collienne C, Roosen J, Ector B, Janssens L, Charlier F, Vankelecom B, Dewilde W, Wijns W. Unifocal Right-Sided Ablation Treatment for Neurally Mediated Syncope and Functional Sinus Node Dysfunction Under Computed Tomographic Guidance. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006604. doi: 10.1161/CIRCEP.118.006604. PMID 30354289
- [Result] Hu F, Zheng L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Right anterior ganglionated plexus: The primary target of cardioneuroablation? Heart Rhythm. 2019 Oct;16(10):1545-1551. doi: 10.1016/j.hrthm.2019.07.018. Epub 2019 Jul 19. PMID 31330187
- [Result] Piotrowski R, Baran J, Kulakowski P. Cardioneuroablation using an anatomical approach: a new and promising method for the treatment of cardioinhibitory neurocardiogenic syncope. Kardiol Pol. 2018;76(12):1736-1738. doi: 10.5603/KP.a2018.0200. Epub 2018 Oct 19. No abstract available. PMID 30338504
- [Result] Oh S, Zhang Y, Bibevski S, Marrouche NF, Natale A, Mazgalev TN. Vagal denervation and atrial fibrillation inducibility: epicardial fat pad ablation does not have long-term effects. Heart Rhythm. 2006 Jun;3(6):701-8. doi: 10.1016/j.hrthm.2006.02.020. Epub 2006 Mar 6. PMID 16731474
- [Result] Pachon M JC, Pachon M EI, Santillana P TG, Lobo TJ, Pachon CTC, Pachon M JC, Albornoz V RN, Zerpa A JC. Simplified Method for Vagal Effect Evaluation in Cardiac Ablation and Electrophysiological Procedures. JACC Clin Electrophysiol. 2015 Oct;1(5):451-460. doi: 10.1016/j.jacep.2015.06.008. Epub 2015 Aug 21. PMID 29759475
- [Result] Romanov A, Minin S, Breault C, Pokushalov E. Visualization and ablation of the autonomic nervous system corresponding to ganglionated plexi guided by D-SPECT 123I-mIBG imaging in patient with paroxysmal atrial fibrillation. Clin Res Cardiol. 2017 Jan;106(1):76-78. doi: 10.1007/s00392-016-1045-2. Epub 2016 Oct 17. No abstract available. PMID 27752762
- [Result] Rose MS, Koshman ML, Ritchie D, Sheldon R. The development and preliminary validation of a scale measuring the impact of syncope on quality of life. Europace. 2009 Oct;11(10):1369-74. doi: 10.1093/europace/eup106. PMID 19797151